CLINICAL TRIAL: NCT02403648
Title: Pharmacokinetics and Pharmacodynamics of BIOD-961 vs. Glucagon for Injection (Eli Lilly) and GlucaGen® (Novo Nordisk) Administered by Subcutaneous and Intramuscular Injection in Normal, Healthy Volunteers
Brief Title: Pharmacokinetics and Pharmacodynamics of BIOD-961 vs. Marketed Glucagons
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biodel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6-101
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Hypoglycemia
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- BIOD-961, 1 mg IM (Experimental): Intramuscular delivery of BIOD-961.
  Interventions: Drug: BIOD-961
- Lilly Glucagon, 1 mg IM (Active Comparator): Intramuscular delivery of Lilly glucagon.
  Interventions: Drug: Lilly Glucagon
- Novo Glucagon, 1 mg IM (Active Comparator): Intramuscular delivery of Novo glucagon.
  Interventions: Drug: Novo Glucagon
- BIOD-961, 1 mg SC (Experimental): Subcutaneous delivery of BIOD-961,
  Interventions: Drug: BIOD-961
- Lilly Glucagon, 1 mg SC (Active Comparator): Subcutaneous delivery of Lilly glucagon.
  Interventions: Drug: Lilly Glucagon
- Novo Glucagon, 1 mg SC (Active Comparator): Subcutaneous delivery of Novo glucagon.
  Interventions: Drug: Novo Glucagon

INTERVENTIONS:
Drug: BIOD-961 — BIOD-961 is a lyophilized glucagon formulation.
  Arms: BIOD-961, 1 mg IM; BIOD-961, 1 mg SC
Drug: Lilly Glucagon
  Arms: Lilly Glucagon, 1 mg IM; Lilly Glucagon, 1 mg SC
Drug: Novo Glucagon
  Arms: Novo Glucagon, 1 mg IM; Novo Glucagon, 1 mg SC

SUMMARY:
BIOD-961 is a dry powder formulation of glucagon intended for use in a device that mixes (reconstitutes) the powder with liquid to make it easier for users to treat patients with severe hypoglycemia. The purpose of this study is to evaluate how much BIOD-961 absorbs into the bloodstream, how much it raises glucose concentrations (the intended effect) and compare to two glucagon products already on the market.

DETAILED DESCRIPTION:
Subjects receive on separate days, in random order one of the following: 1 mg BIOD-961 intramuscularly (IM), 1 mg Lilly (IM), 1 mg Novo (IM), 1 mg BIOD-961 subcutaneously (SC), 1 mg Lilly (SC), and 1 mg Novo (SC).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index: 18.5-25.0 kg/m2 inclusive.
* Subject has provided informed consent and has signed and dated an informed consent form before any trial-related activities.

Exclusion Criteria:

* Type 1 or type 2 diabetes mellitus.
* History of pheochromocytoma, insulinoma, glucagonoma, or glycogen storage disease.
* History of regular alcohol consumption as defined by alcohol intake exceeding 7 drinks per week for females or 14 drinks per week for males, where 1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor.
* Significant cardiovascular (to include New York Heart Association (NYHA) Class III or- IV functional capacity or uncontrolled hypertension), respiratory, gastrointestinal, hepatic, renal, neurological, psychiatric and/or hematological disease.
* Any significant cardiovascular event history, including angina, myocardial infarction, therapeutic coronary procedure (e.g, percutaneous transluminal coronary angioplasty, coronary bypass surgery), stroke, or transient ischemic attack.
* Females who are breast feeding, pregnant, or intending to become pregnant during the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Glucagon maximal concentration and area under curve | 240 minutes post dose
Glucose maximal concentration and area under curve | 240 minutes after dose

SECONDARY OUTCOMES:
Time to maximal glucagon concentration | 240 minutes after dose
Time to maximal glucose concentration | 240 minutes after dose
Maximal glucose excursion | 240 minutes after dose
Area under the glucose time curve from 0 to return to baseline after blood glucose peaked | 240 minutes after dose

CONTACTS AND LOCATIONS:
Overall Officials: Linda Morrow, MD, Principal Investigator — Profil Institute for Clinical Research, Inc.; Alan Krasner, MD, Study Director — Biodel